CLINICAL TRIAL: NCT02194361
Title: Efficacy of a Bilberry Extract Standardised to a Content of 25% Anthocyanosides in Improving the Night Vision of Healthy Volunteers: a Double-blind, Randomized, Placebo Controlled, Cross-over Trial Over 2 x 28 Days
Brief Title: Efficacy of a Standardised Bilberry Extract in Improving the Night Vision of Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1147.3
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Anthocyan capsules (Experimental)
  Interventions: Drug: Anthocyan capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anthocyan capsules — Bilberry extract capsules, 160 mg (25% anthocyanosides)
  Arms: Anthocyan capsules
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to determine the Efficacy of Standardised Bilberry Extract in improving the night vision and to evaluate its tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (volunteers) with normal twilight and night vision
* Age 18+, young and collaborative men or women
* Having given their written informed consent
* Full visual acuity (vision 0.8 or better) according to DIN Standard condition
* Refraction ≤ +/-10.0 in the highest main step
* Normal intraocular pressure (10-20 mmHg)

Exclusion Criteria:

* Diabetes mellitus
* Epilepsy
* Abnormal visual acuity or abnormal morphological eye findings
* Glaucoma and macula degeneration
* Disease of the retina
* Consumption of anthocyan preparations during the past six months
* Opthalmologic pathology: cataract, visus < 0.8, retinal pathology, maculopathy, intraocular pressure > 21 mmHg, known acute or chronic eye disease, use of hard contact lenses, eye surgery performed within the last 12 months
* Any serious disorder that might interfere with his/her participation in this study and the evaluation of the efficacy or safety of the test drug: e.g. diabetes mellitus, anamnestic indications of diabetic microangiopathy or polyneuropathy, renal insufficiency, hepatic or metabolic dysfunction, cardiovascular disease (hypertension > 160/100 mmHg), psychiatric disorder, myasthenia gravis, delirious state, albino
* Any treatment that might interfere with the evaluation of the test drug, in particular drugs with known influence on eye sight or adaptation (e.g. chloroquine, digitalis, ethambutol, chlorpromazine, benzodiazepines or phenothiazine derivatives such as thioridazine, periciazine, perphenazine)
* Known hypersensitivity to any of the ingredients of the study drug
* Drug and alcohol abuse
* Pregnancy, lactation, women of childbearing potential who do not use an established contraceptive
* Participation in another trial within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 1999-12; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Change of the dark adaption of the pupil using the method of the dark adaption Goggles (DAG) | From day 1 to 28 and from day 57 to day 84

SECONDARY OUTCOMES:
Changes of the dark adaption using dark flashes | From day 1 to day 28 and from day 57 to day 84
  Pupillography (PG)
Changes of the weakest, correctly recognised contrast level | From day 1 to day 28 and from day 57 to day 84
  Mesoptometry
Assessment of subjective efficacy based on a visual analogue scale (VAS) rating questionnaire | pre-dose on day 1, day 28, pre-dose on day 57, day 84
Assessment of clinical global impression on a 5-point rating scale | Days 28 and 84